CLINICAL TRIAL: NCT03165812
Title: Single Anastomosis Duodeno Jejunal Bypass With Sleeve Gastrectomy (SADJB-SG) Versus Intensive Medical Therapy (IMT) in the Treatment of Type 2 Diabetes Mellitus Among Asian Patients With BMI 23.5 - 30 kg/m2: A Clinical Trial
Brief Title: A Diabetes Improvement in Medical Therapy Versus SADJB Study
Acronym: DIMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Tikfu Gee, Senior lecturer/ consultant, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-16-1486-32126
Record Dates: First submitted 2017-04-14; First posted 2017-05-24 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 2; Overweight
Keywords: Sleeve Gastrectomy; Duodeno Jejunal Bypass; Single Anastomosis; Intensive Medical Therapy; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study will involve two groups with equal allocation of patients in the intensive medical therapy (IMT) group and Single Anastomosis Duodeno Jejunal Bypass with Sleeve Gastrectomy (SADJB-SG) group with stratification by use of insulin at screening. All patients who agree to participate in this study will be assigned to one of the treatment groups by the doctor without randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SADJB-SG group (Experimental): Patients in this group will undergo bariatric surgery. There are two parts to this procedure. One is the restrictive type of weight loss surgery, which reduces the stomach size. The other type prevents the body from absorbing fats and sugar properly, as the small intestine will be attached to the small stomach, bypassing most of the stomach and upper part of the small intestine. This surgery will be performed using a minimally invasive technique known as laparoscopic keyhole surgery.
  Interventions: Procedure: SADJB-SG group
- IMT group (Experimental): Patients in this group will be subjected to strict adherence to diet, optimisation of diabetic medications and close monitoring of blood glucose and HbA1c.
  Interventions: Procedure: IMT group

INTERVENTIONS:
Procedure: SADJB-SG group — Patients will undergo bariatric surgery. A clear liquid high protein diet will be started in the first two postoperative days. If no complications were detected by physical examination, patients will be stimulated to walk and will be dismissed from the hospital on postoperative day 3. Patients will be subjected to a strict adherence to diet and close monitoring of their blood glucose and HbA1c levels during the study period. Standard follow-up includes a visit to the outpatient clinic at 1, 2, 3, 4 weeks after surgery, then 3, 6, 9, 12, 18, 24 months and after that, a life-long annual visit. Glycaemic control at home will be maintained as in the preoperative period and patients will need to inform the results of their blood glucose levels to the doctor during each follow-up visits.
  Arms: SADJB-SG group
Procedure: IMT group — Patients will be subjected to strict adherence to their diet, optimisation of their diabetic medications and close monitoring of their blood glucose and HbA1c levels at 0, 6, 12, 24 months. The endocrinologist will be monitoring the patients in this group. Detailed individualized lifestyle and dietary counseling will be given by a dietitian emphasizing on nutrition knowledge, the timing of meal with medication, portion control, and increasing daily physical activity level.
  Arms: IMT group

SUMMARY:
The incidence of diabetes mellitus is increasing annually in Asia. It is the leading cause of blindness, chronic renal insufficiency, and amputations, multiplying the risks of heart disease and stroke. Ninety percent of diabetic patients are type 2 diabetes mellitus (T2DM), which is usually associated with overweight and obese. Single Anastomosis Duodeno-Jejunal Bypass with Sleeve Gastrectomy (SADJB-SG) is a type of bariatric surgery whereby food is bypassed into the distal jejunum, and the duodenum is excluded. Sleeve gastrectomy offers the restrictive component by reducing the capacity of the stomach. In short, this combined technique results in food restriction and malabsorption. A total of 84 patients will be recruited in this study. An equal number of patients will be allocated into two groups. There will be an intensive medical therapy group (IMT) and SADJB-SG group. The patients in IMT group will be subjected to strict adherence to diet, optimization of diabetic medications and close monitoring of blood glucose and glycated haemoglobin (HbA1c) level. The SADJB-SG group will be undergoing surgery. The variables that will be studied include body mass index (BMI), fasting blood glucose (FBG), glycated haemoglobin (HbA1c), C- peptide, plasma insulin and Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). Biochemical markers are important in this research as the development of T2DM involves both multi-organ insulin resistance and inadequate insulin secretion by pancreatic β-cells, leading to high blood sugar during fasting and post meal. Other mechanisms proposed in this study are leptin, adipokines, incretins, amino acids, and diabetic dyslipidaemia. The raw data will be analysed using the SPSS statistical software. At the end of the study, the investigator will evaluate and determine the role of SADJB-SG in glycaemic control and BMI in T2DM patients compared to IMT. The investigator hypothesized that there is an improvement in HbA1c level in T2DM patients in SADJB-SG group compare to IMT group.

DETAILED DESCRIPTION:
Recruitment will be a prospective study in patients with body mass index (BMI) of 23.5-30 kg/m2, aged between 18 and 65 years old. Each patient will be preoperatively screened (including psychologist assessment) and evaluated by the study multidisciplinary team before recruitment. The study will involve two groups with equal allocation of patients in the intensive medical therapy (IMT) group and Single Anastomosis Duodeno Jejunal Bypass with Sleeve Gastrectomy (SADJB-SG) group with stratification by use of insulin at screening. All patients who agree to participate in this study will be assigned to one of the treatment groups by the doctor without randomization. Before making a final decision for treatment, every patient will undergo a detailed and up-to-date evaluation by the doctor regarding the suitability, the pros and cons, risk and benefits, the potential postoperative complications and the likelihood of requiring postoperative nutritional supplementation. Patients that are eligible to take part in this study will be informed, and the final decision will solely be made based on patients' willingness. The patients will also be made aware that this is an experimental trial and both verbal and written informed consent will be taken before treatment. In addition, the patients will be informed regarding the use of the clinical and analytical data for publication purposes. Initial assessment of the patient's social demographic data, history of present illness (duration of diabetes, oral hypoglycemic agent used), medical and surgical history, family history, anthropometric measurements (height, weight, BMI, calculated as weight (kg)/height (m2), waist, hip and neck circumference), history of weight loss attempt, diet and lifestyle assessment, quality of life assessment and biochemical measures including fasting blood glucose (FBG), glycated haemoglobin (HbA1c), C- peptide, plasma insulin and HOMA-IR, assessment for obstructive sleep apnea, depression and sleep quality will be obtained upon approval of participation in the study or before any form of treatment. An additional pre-operation questionnaire will be given to the SADJB-SG group during initial assessment to ensure understanding of the patients towards the surgery. Adverse events will be monitored closely at 1, 2, 3, and 4 weeks after surgery. In any occurrence of an adverse event, it will be documented and reported within 14 days.The study will be terminated if there are life-threatening or severe adverse events associated with SADJB-SG group or IMT group.

Patients will not be given access to the study data however the patients will be informed regarding their progress during every follow-up visit. All medical records and research data will be kept in the investigator's hard disk and web-based storage (i-cloud and i-drive) for two years. Study data will be held even after the study period as there will still be a continuous follow-up with the patients for life. However, all patients' information obtained from this study will be kept and handled in a confidential manner, by applicable laws and regulations. When publishing or presenting the study results, the identity of patients will not be revealed without patient's expressed consent. Participants will also be covered under clinical trial insurance from the institution during the study period. In the case of emergency, all patients will be given the contact number of the investigator as the investigators are contactable throughout the day. This study will begin after receiving the approval of Medical Research & Ethics Committee, Ministry of Health Malaysia.

Sample size:

The sample size was estimated with the help of PS software (power and sample size calculation software) 3.1.2 with a power of 80% and a significant level of 0.05. The estimation was based on the diabetic remission in a few study done on bariatric surgery on one arm and intensive medical treatment on the other and it was detected a range of 57% to 73% diabetic remission among the bariatric surgery group. Another study by Lee WJ et al., 2014 found a diabetic remission rate of 64% (HbA1C<6.0%) with the SADJB-SG group one year after surgery. The total estimated sample size is 34 patients in each arm for this study. However, with the inclusion of 20% dropout rate, the total number of patients needed for this study is 42 patients in each arm.

Laboratory investigations:

15 ml of fasting blood samples will be taken early in the morning for the following blood tests stated below in Ethylenediaminetetraacetic acid (EDTA), fluoride oxalate and plain tubes, depending on the respective test. Samples will be further centrifuged for the serum to be stored in 3 aliquots (1 ml each) for batch analysis. This serum will be stored at - 80°C pending further analysis. The analysis will be done at the Chemical Pathology Laboratory, Faculty of Medicine & Health Sciences, UPM.3.6.1. Baseline preoperative biochemical markers and profiles for all bariatric surgery T2DM candidates, and other nutrients 'at risk' related to medication usage or poor dietary quality include:

Blood investigations on automated analyser:

* Full blood count
* Renal profile (urea, creatinine, sodium, potassium)
* Liver function test (total protein, albumin, bilirubin, alkaline phosphatase, alanine transaminase, aspartate aminotransferase, gamma-glutamyl transferase)
* Thyroid function test (TSH, free T4)
* Cortisol
* Fasting plasma glucose, HbA1c
* Fasting lipid profile (total cholesterol, triglyceride, LDL, HDL)
* Bone profile [calcium, phosphate, magnesium, parathyroid hormone, 25-OH vitamin D]
* Iron, ferritin, vitamin B12, folate

Urine investigations

* Urinalysis (dipstick) & urine FEME (automated analyser)
* Urine microalbumin (automated analyser)

These investigations will be repeated in 24 months but more frequently if clinically indicated. Apart from that, studying the following parameters at baseline, 6 and 12 months post-surgery will allow us to explore the hypothesis that a modulatory effect on incretin production could lead to better glycaemic control independent of weight loss.

* Insulin, C-peptide (automated analyser), HOMA-IR (calculated value)
* Lipoprotein Subfractionation on Lipoprint LDL system.
* Incretins (GLP-1, GIP)
* Adipokines such as leptin
* Adiponectin
* FGF19 (Fibroblast Growth Factor 19)
* Tumor necrosis factor-alpha (TNF-alpha)

Genetic Analysis:

DNA Extraction- Laboratory analyses will be obtained after an overnight fast and the plasma will be separated by centrifugation and storage at -20ºC. The available commercial DNA extraction methods will be utilized to get a good DNA regarding quantity and quality.

DNA Quantification- The quality of the extracted DNA will be evaluated using electrophoresis and the concentration of the extracted DNA will be estimated using the spectrophotometer.

Genotyping analysis-

* Standardization of Polymerase chain reaction (PCR) will be carried out for the respective genes.
* Identification and analysis of candidate genes polymorphisms of GCG, GLP1R, DPP4, GIP, GIPR and PCSK1 genes by conventional PCR, PCR-RFLP, Real time- PCR High Resolution Analysis.

Staining and Visualizing of Genomic DNA- Agarose electrophoresis will be carried out to determine the PCR products by staining with ethidium bromide. The genomic DNA, PCR amplified products and the restricted fragments will be visualized under ultraviolet light and the image will be captured by Alpha Imager.

Validation- Nearly 10% of the samples will be randomly chosen and the samples will be genotyped on the same assay for the second time and the results will be scored by the other researcher.

Positive and Negative Controls PCR amplified products from the respective gene will be sequenced to identify the genotypes. Those samples will be used as a positive control for the respective genes and the PCR grade water lacking the DNA template will be used as a negative control.

DNA Sequencing methods-

* DNA sequencing will be done to confirm the polymorphism of the respective genes.
* The sequencing results will be subjected to BLAST (www.ncbi.nlm.nig.gov/BLAST) and it has been verified against the published gene sequence for the respective gene.

Data Analysis:

Statistical calculations will be performed using the standard statistical software package, IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp. Results will be expressed as mean values and standard deviation for normally distributed variables. Median and interquartile range (IQR) will be calculated for all not normally distributed continuous variables. Non-parametric tests such as Mann-Whitney U test and/or Kruskall-Wallis test will be used for non-normal distribution of variables. Associations between qualitative variables will be determined by Chi-square test, Fisher's exact test and SAS Exact Contingency Table. In all statistical analyses, p-value of < 0.05 (95% confidence interval) was considered to be statistically significant.

Analysis of variance (ANOVA) will be used to test for significant differences between means.

* Univariate logistic regression analysis will be used to determine the synergistic effect of the genetic variants
* The Hardy-Weinberg equilibrium for genotypic distribution will be evaluated using the Hardy-Weinberg equilibrium exact test.
* Rotor-Gene 6000 software (software version 1.7, built 87) will be used for the HRM analysis for certain gene polymorphisms by generating a normalized melting curve, a difference graph and a derivative plot.

The categorical variables from this study such as Body Mass Index (BMI), fasting glucose, HbA1c, C- peptide levels, Plasma insulin and HOMA-IR will be reported as counts and percent and compared between SADJB-SG group and IMT group by SPSS method.

Study Ethics:

Ethical clearance will be obtained from the Ethics Committee for Research Involving Human Subjects Universiti Putra Malaysia (JKEUPM) and Kuala Lumpur General Hospital. This study will be submitted to National Medical Research Register (NMRR) for Medical Research and Ethics Committee, Ministry of Health Malaysia (MREC) clearance. Informed consent will be obtained from each participant of the study.

Conflict of Interest:

There is no conflict of interest among the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* BMI 23.5 - 30 kg/m2.
* Diabetes more than two years and less than ten years.
* American Society of Anesthesiologists (ASA) classification < 4
* Able to give informed consent

Exclusion Criteria:

* Age: below 18 and above 65.
* Inability to informed consent.
* Patients on GLP-1 agonist and insulin two weeks before admission into the trial.
* Diabetes more than ten years or less than two years.
* C-Peptide level < 2.0 ng/mL
* American Society of Anesthesiologists (ASA) classification > 3
* Logistic issue where patient come from rural area and has difficulty in complying with the post-operation close monitoring and follow-up
* Patient who has psychiatric disorder (depression, substance abuse, eating disorder, alcoholism, dementia etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Type 2 Diabetes Mellitus (T2DM) patients in SADJB-SG group achieving glycated hemoglobin (HbA1c) level of less than 7% (with or without diabetes medications) in 2 years as compare to patients in IMT group. | 24 months
  The HbA1c level is measured in percentage

SECONDARY OUTCOMES:
T2DM patients in SADJB-SG group achieving mean fasting blood glucose level of 4.4-7.0 mmol/l in 2 years as compare to patients in IMT group. | 24 months
  Fasting blood glucose level is measured in mmol/l
T2DM patients in SADJB-SG group achieving lower body mass index (BMI) in 2 years as compare to IMT group. | 24 months
  BMI is calculated as weight (kg)/height (m^2)
Changes in serum level of lipids. | 24 months
  Fasting blood samples will be taken early in the morning. In the study, serum concentrations of the following lipids will be measured using automated clinical chemistry analyzer: triglycerides, total cholesterol, HDL, LDL. LDL-Subfractionation will be done using Quantrimetrix Lipoprint system. The measurements will be performed before the planned intervention and then at intervals of 6, 12 and 24 months. The results will be presented in respective units (mmol/L).
Assessment of NAFLD associated morbidities by detecting the metabolic changes after SADJB-SG. | 24 months
  In the study, serum concentrations of the following analytes will be measured on an automated clinical chemistry analyzer: total protein (g/L), albumin (g/L), bilirubin (umol/L), alkaline phosphatase (U/L), alanine transaminase (U/L), aspartate aminotransferase (U/L), gamma-glutamyl transferase (U/L). ELISA Technique will be used to analyze the following parameters in serum: leptin (pg/mL), adiponectin, FGF19 (pg/mL), and TNF-alpha (pg/mL). The measurements will be performed before the planned intervention and then at intervals of 6, 12 and 24 months.
Identification of proposed mechanism for improvement in glycemic control following SADJB-SG. | 24 months
  In the study, serum incretins GLP-1 (pmol/L) and GIP (pmol/L) will be analyzed using ELISA technique. The measurements will be performed before the planned intervention and then at intervals of 6, 12 and 24 months.
Identification of genetic biomarkers. | Baseline
  The genotypic and allelic frequencies of genetic polymorphisms of GCG, GLP1R, DPP4, GIP, GIPR, PCSK1 gene are analyzed by PCR method. The significant association (p<0.05) of genetic polymorphisms between the subjects is considered as the genetic risk factors/genetic marker for the development of T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Tikfu Gee, MBBS, MS, Principal Investigator — Universiti Putra Malaysia
Locations (2):
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital Serdang, Kajang, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmet P, Alberti KG, Shaw J. Global and societal implications of the diabetes epidemic. Nature. 2001 Dec 13;414(6865):782-7. doi: 10.1038/414782a. PMID 11742409
- [Background] Greenway SE, Greenway FL 3rd, Klein S. Effects of obesity surgery on non-insulin-dependent diabetes mellitus. Arch Surg. 2002 Oct;137(10):1109-17. doi: 10.1001/archsurg.137.10.1109. PMID 12361414
- [Background] Guh DP, Zhang W, Bansback N, Amarsi Z, Birmingham CL, Anis AH. The incidence of co-morbidities related to obesity and overweight: a systematic review and meta-analysis. BMC Public Health. 2009 Mar 25;9:88. doi: 10.1186/1471-2458-9-88. PMID 19320986
- [Background] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Background] Bradley D, Magkos F, Klein S. Effects of bariatric surgery on glucose homeostasis and type 2 diabetes. Gastroenterology. 2012 Oct;143(4):897-912. doi: 10.1053/j.gastro.2012.07.114. Epub 2012 Aug 8. PMID 22885332
- [Background] Pories WJ, MacDonald KG Jr, Flickinger EG, Dohm GL, Sinha MK, Barakat HA, May HJ, Khazanie P, Swanson MS, Morgan E, et al. Is type II diabetes mellitus (NIDDM) a surgical disease? Ann Surg. 1992 Jun;215(6):633-42; discussion 643. doi: 10.1097/00000658-199206000-00010. PMID 1632685
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Lee WJ, Huang MT, Wang W, Lin CM, Chen TC, Lai IR. Effects of obesity surgery on the metabolic syndrome. Arch Surg. 2004 Oct;139(10):1088-92. doi: 10.1001/archsurg.139.10.1088. PMID 15492149
- [Background] Madan AK, Orth W, Ternovits CA, Tichansky DS. Metabolic syndrome: yet another co-morbidity gastric bypass helps cure. Surg Obes Relat Dis. 2006 Jan-Feb;2(1):48-51; discussion 51. doi: 10.1016/j.soard.2005.09.014. PMID 16925317
- [Background] Mottin CC, Vontobel Padoin A, Schroer CE, Barancelli FT, Glock L, Repetto G. Behavior of type 2 diabetes mellitus in morbid obese patients submitted to gastric bypass. Obes Surg. 2008 Feb;18(2):179-81. doi: 10.1007/s11695-007-9249-1. Epub 2008 Jan 4. PMID 18176858
- [Background] Rubino F, Marescaux J. Effect of duodenal-jejunal exclusion in a non-obese animal model of type 2 diabetes: a new perspective for an old disease. Ann Surg. 2004 Jan;239(1):1-11. doi: 10.1097/01.sla.0000102989.54824.fc. PMID 14685093
- [Background] Rubino F, Forgione A, Cummings DE, Vix M, Gnuli D, Mingrone G, Castagneto M, Marescaux J. The mechanism of diabetes control after gastrointestinal bypass surgery reveals a role of the proximal small intestine in the pathophysiology of type 2 diabetes. Ann Surg. 2006 Nov;244(5):741-9. doi: 10.1097/01.sla.0000224726.61448.1b. PMID 17060767
- [Background] Dixon JB, O'Brien PE, Playfair J, Chapman L, Schachter LM, Skinner S, Proietto J, Bailey M, Anderson M. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA. 2008 Jan 23;299(3):316-23. doi: 10.1001/jama.299.3.316. PMID 18212316
- [Background] O'Brien PE, Dixon JB, Laurie C, Skinner S, Proietto J, McNeil J, Strauss B, Marks S, Schachter L, Chapman L, Anderson M. Treatment of mild to moderate obesity with laparoscopic adjustable gastric banding or an intensive medical program: a randomized trial. Ann Intern Med. 2006 May 2;144(9):625-33. doi: 10.7326/0003-4819-144-9-200605020-00005. PMID 16670131
- [Background] Corsini DA, Simoneti CA, Moreira G, Lima SE Jr, Garrido AB. Cancer in the excluded stomach 4 years after gastric bypass. Obes Surg. 2006 Jul;16(7):932-4. doi: 10.1381/096089206777822313. PMID 16839497
- [Background] Harper JL, Beech D, Tichansky DS, Madan AK. Cancer in the bypassed stomach presenting early after gastric bypass. Obes Surg. 2007 Sep;17(9):1268-71. doi: 10.1007/s11695-007-9216-x. PMID 18074505
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Background] Lovshin JA, Drucker DJ. Incretin-based therapies for type 2 diabetes mellitus. Nat Rev Endocrinol. 2009 May;5(5):262-9. doi: 10.1038/nrendo.2009.48. PMID 19444259
- [Result] Cohen RV, Neto MG, Correa JL, Sakai P, Martins B, Schiavon CA, Petry T, Salles JE, Mamedio C, Sorli C. A pilot study of the duodenal-jejunal bypass liner in low body mass index type 2 diabetes. J Clin Endocrinol Metab. 2013 Feb;98(2):E279-82. doi: 10.1210/jc.2012-2814. Epub 2013 Jan 21. PMID 23337729
- [Result] Cohen R, Pinheiro JS, Correa JL, Schiavon CA. Laparoscopic Roux-en-Y gastric bypass for BMI < 35 kg/m(2): a tailored approach. Surg Obes Relat Dis. 2006 May-Jun;2(3):401-4, discussion 404. doi: 10.1016/j.soard.2006.02.011. PMID 16925363
- [Result] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric surgery versus intensive medical therapy for diabetes--3-year outcomes. N Engl J Med. 2014 May 22;370(21):2002-13. doi: 10.1056/NEJMoa1401329. Epub 2014 Mar 31. PMID 24679060
- [Result] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Result] Lee WJ, Chong K, Ser KH, Lee YC, Chen SC, Chen JC, Tsai MH, Chuang LM. Gastric bypass vs sleeve gastrectomy for type 2 diabetes mellitus: a randomized controlled trial. Arch Surg. 2011 Feb;146(2):143-8. doi: 10.1001/archsurg.2010.326. PMID 21339423
- [Result] Lee WJ, Lee KT, Kasama K, Seiki Y, Ser KH, Chun SC, Chen JC, Lee YC. Laparoscopic single-anastomosis duodenal-jejunal bypass with sleeve gastrectomy (SADJB-SG): short-term result and comparison with gastric bypass. Obes Surg. 2014 Jan;24(1):109-13. doi: 10.1007/s11695-013-1067-z. PMID 23990452
- [Result] Sanchez-Pernaute A, Herrera MA, Perez-Aguirre ME, Talavera P, Cabrerizo L, Matia P, Diez-Valladares L, Barabash A, Martin-Antona E, Garcia-Botella A, Garcia-Almenta EM, Torres A. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S). One to three-year follow-up. Obes Surg. 2010 Dec;20(12):1720-6. doi: 10.1007/s11695-010-0247-3. PMID 20798995
- [Result] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Result] Lee WJ, Almulaifi AM, Tsou JJ, Ser KH, Lee YC, Chen SC. Duodenal-jejunal bypass with sleeve gastrectomy versus the sleeve gastrectomy procedure alone: the role of duodenal exclusion. Surg Obes Relat Dis. 2015 Jul-Aug;11(4):765-70. doi: 10.1016/j.soard.2014.12.017. Epub 2014 Dec 24. PMID 25813754
- [Result] Garcia-Caballero M, Valle M, Martinez-Moreno JM, Miralles F, Toval JA, Mata JM, Osorio D, Minguez A. Resolution of diabetes mellitus and metabolic syndrome in normal weight 24-29 BMI patients with One Anastomosis Gastric Bypass. Nutr Hosp. 2012 Mar-Apr;27(2):623-31. doi: 10.1590/S0212-16112012000200041. PMID 22732993
- [Result] Bose M, Olivan B, Teixeira J, Pi-Sunyer FX, Laferrere B. Do Incretins play a role in the remission of type 2 diabetes after gastric bypass surgery: What are the evidence? Obes Surg. 2009 Feb;19(2):217-229. doi: 10.1007/s11695-008-9696-3. Epub 2008 Sep 27. PMID 18820978
- [Result] Laferrere B. Diabetes remission after bariatric surgery: is it just the incretins? Int J Obes (Lond). 2011 Sep;35 Suppl 3(0 3):S22-5. doi: 10.1038/ijo.2011.143. PMID 21912382
- [Result] Chronaiou A, Tsoli M, Kehagias I, Leotsinidis M, Kalfarentzos F, Alexandrides TK. Lower ghrelin levels and exaggerated postprandial peptide-YY, glucagon-like peptide-1, and insulin responses, after gastric fundus resection, in patients undergoing Roux-en-Y gastric bypass: a randomized clinical trial. Obes Surg. 2012 Nov;22(11):1761-70. doi: 10.1007/s11695-012-0738-5. PMID 22911148
- [Result] Geloneze B, Geloneze SR, Chaim E, Hirsch FF, Felici AC, Lambert G, Tambascia MA, Pareja JC. Metabolic surgery for non-obese type 2 diabetes: incretins, adipocytokines, and insulin secretion/resistance changes in a 1-year interventional clinical controlled study. Ann Surg. 2012 Jul;256(1):72-8. doi: 10.1097/SLA.0b013e3182592c62. PMID 22664560
- [Result] Goktas Z, Moustaid-Moussa N, Shen CL, Boylan M, Mo H, Wang S. Effects of bariatric surgery on adipokine-induced inflammation and insulin resistance. Front Endocrinol (Lausanne). 2013 Jun 10;4:69. doi: 10.3389/fendo.2013.00069. eCollection 2013. PMID 23772224
- [Result] Enkhmaa B, Shiwaku K, Anuurad E, Nogi A, Kitajima K, Yamasaki M, Oyunsuren T, Yamane Y. Prevalence of the metabolic syndrome using the Third Report of the National Cholesterol Educational Program Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (ATP III) and the modified ATP III definitions for Japanese and Mongolians. Clin Chim Acta. 2005 Feb;352(1-2):105-13. doi: 10.1016/j.cccn.2004.08.012. PMID 15653104
- [Result] Pyorala K, Pedersen TR, Kjekshus J, Faergeman O, Olsson AG, Thorgeirsson G. Cholesterol lowering with simvastatin improves prognosis of diabetic patients with coronary heart disease. A subgroup analysis of the Scandinavian Simvastatin Survival Study (4S). Diabetes Care. 1997 Apr;20(4):614-20. doi: 10.2337/diacare.20.4.614. PMID 9096989
- [Result] Foger B. Lipid lowering therapy in type 2 diabetes. Wien Med Wochenschr. 2011 Jun;161(11-12):289-96. doi: 10.1007/s10354-011-0908-4. PMID 21769710
- [Result] Inukai T, Yamamoto R, Suetsugu M, Matsumoto S, Wakabayashi S, Inukai Y, Matsutomo R, Takebayashi K, Aso Y. Small low-density lipoprotein and small low-density lipoprotein/total low-density lipoprotein are closely associated with intima-media thickness of the carotid artery in Type 2 diabetic patients. J Diabetes Complications. 2005 Sep-Oct;19(5):269-75. doi: 10.1016/j.jdiacomp.2005.03.002. PMID 16112502
- [Result] Superko HR, Gadesam RR. Is it LDL particle size or number that correlates with risk for cardiovascular disease? Curr Atheroscler Rep. 2008 Oct;10(5):377-85. doi: 10.1007/s11883-008-0059-2. PMID 18706278
- [Result] Syvanne M, Ahola M, Lahdenpera S, Kahri J, Kuusi T, Virtanen KS, Taskinen MR. High density lipoprotein subfractions in non-insulin-dependent diabetes mellitus and coronary artery disease. J Lipid Res. 1995 Mar;36(3):573-82. PMID 7775869
- [Result] Asztalos BF, Cupples LA, Demissie S, Horvath KV, Cox CE, Batista MC, Schaefer EJ. High-density lipoprotein subpopulation profile and coronary heart disease prevalence in male participants of the Framingham Offspring Study. Arterioscler Thromb Vasc Biol. 2004 Nov;24(11):2181-7. doi: 10.1161/01.ATV.0000146325.93749.a8. Epub 2004 Sep 23. PMID 15388521
- [Result] Soran H, Hama S, Yadav R, Durrington PN. HDL functionality. Curr Opin Lipidol. 2012 Aug;23(4):353-66. doi: 10.1097/MOL.0b013e328355ca25. PMID 22732521
- [Result] Krauss RM, Siri PW. Metabolic abnormalities: triglyceride and low-density lipoprotein. Endocrinol Metab Clin North Am. 2004 Jun;33(2):405-15. doi: 10.1016/j.ecl.2004.03.016. PMID 15158526
- [Result] Nassif AT, Nagano TA, Okayama S, Nassif LS, Branco Filho A, Sampaio Neto J. Performance of the Bard Scoring System in Bariatric Surgery Patients with Nonalcoholic Fatty Liver Disease. Obes Surg. 2017 Feb;27(2):394-398. doi: 10.1007/s11695-016-2284-z. PMID 27392972
- [Result] Frantzides CT, Carlson MA, Moore RE, Zografakis JG, Madan AK, Puumala S, Keshavarzian A. Effect of body mass index on nonalcoholic fatty liver disease in patients undergoing minimally invasive bariatric surgery. J Gastrointest Surg. 2004 Nov;8(7):849-55. doi: 10.1016/j.gassur.2004.07.001. PMID 15531238
- [Result] Taitano AA, Markow M, Finan JE, Wheeler DE, Gonzalvo JP, Murr MM. Bariatric surgery improves histological features of nonalcoholic fatty liver disease and liver fibrosis. J Gastrointest Surg. 2015 Mar;19(3):429-36; discussion 436-7. doi: 10.1007/s11605-014-2678-y. Epub 2014 Dec 24. PMID 25537957
- [Result] Furuya CK Jr, de Oliveira CP, de Mello ES, Faintuch J, Raskovski A, Matsuda M, Vezozzo DC, Halpern A, Garrido AB Jr, Alves VA, Carrilho FJ. Effects of bariatric surgery on nonalcoholic fatty liver disease: preliminary findings after 2 years. J Gastroenterol Hepatol. 2007 Apr;22(4):510-4. doi: 10.1111/j.1440-1746.2007.04833.x. PMID 17376042
- [Result] van Dijk SJ, Molloy PL, Varinli H, Morrison JL, Muhlhausler BS; Members of EpiSCOPE. Epigenetics and human obesity. Int J Obes (Lond). 2015 Jan;39(1):85-97. doi: 10.1038/ijo.2014.34. Epub 2014 Feb 25. PMID 24566855
- [Result] Prasadan K, Koizumi M, Tulachan S, Shiota C, Lath N, Paredes J, Guo P, El-Gohary Y, Malek M, Shah S, Gittes GK. The expression and function of glucose-dependent insulinotropic polypeptide in the embryonic mouse pancreas. Diabetes. 2011 Feb;60(2):548-54. doi: 10.2337/db09-0035. PMID 21270265
- [Result] Miyawaki K, Yamada Y, Ban N, Ihara Y, Tsukiyama K, Zhou H, Fujimoto S, Oku A, Tsuda K, Toyokuni S, Hiai H, Mizunoya W, Fushiki T, Holst JJ, Makino M, Tashita A, Kobara Y, Tsubamoto Y, Jinnouchi T, Jomori T, Seino Y. Inhibition of gastric inhibitory polypeptide signaling prevents obesity. Nat Med. 2002 Jul;8(7):738-42. doi: 10.1038/nm727. Epub 2002 Jun 17. PMID 12068290
- [Result] Choquet H, Kasberger J, Hamidovic A, Jorgenson E. Contribution of common PCSK1 genetic variants to obesity in 8,359 subjects from multi-ethnic American population. PLoS One. 2013;8(2):e57857. doi: 10.1371/journal.pone.0057857. Epub 2013 Feb 25. PMID 23451278
- [Result] Chang YC, Chiu YF, Shih KC, Lin MW, Sheu WH, Donlon T, Curb JD, Jou YS, Chang TJ, Li HY, Chuang LM. Common PCSK1 haplotypes are associated with obesity in the Chinese population. Obesity (Silver Spring). 2010 Jul;18(7):1404-9. doi: 10.1038/oby.2009.390. Epub 2009 Oct 29. PMID 19875984
- [Result] Heo YS, Park JM, Kim YJ, Kim SM, Park DJ, Lee SK, Han SM, Shim KW, Lee YJ, Lee JY, Kwon JW. Bariatric surgery versus conventional therapy in obese Korea patients: a multicenter retrospective cohort study. J Korean Surg Soc. 2012 Dec;83(6):335-42. doi: 10.4174/jkss.2012.83.6.335. Epub 2012 Nov 27. PMID 23230551
- [Result] Cummings DE, Arterburn DE, Westbrook EO, Kuzma JN, Stewart SD, Chan CP, Bock SN, Landers JT, Kratz M, Foster-Schubert KE, Flum DR. Gastric bypass surgery vs intensive lifestyle and medical intervention for type 2 diabetes: the CROSSROADS randomised controlled trial. Diabetologia. 2016 May;59(5):945-53. doi: 10.1007/s00125-016-3903-x. Epub 2016 Mar 17. PMID 26983924
- [Result] Ikramuddin S, Korner J, Lee WJ, Bantle JP, Thomas AJ, Connett JE, Leslie DB, Inabnet WB 3rd, Wang Q, Jeffery RW, Chong K, Chuang LM, Jensen MD, Vella A, Ahmed L, Belani K, Olofson AE, Bainbridge HA, Billington CJ. Durability of Addition of Roux-en-Y Gastric Bypass to Lifestyle Intervention and Medical Management in Achieving Primary Treatment Goals for Uncontrolled Type 2 Diabetes in Mild to Moderate Obesity: A Randomized Control Trial. Diabetes Care. 2016 Sep;39(9):1510-8. doi: 10.2337/dc15-2481. Epub 2016 Jun 16. PMID 27311493